CLINICAL TRIAL: NCT04440423
Title: Bioavailability of a Formulation of Clotiazepam 5 mg Coated Tablets With Regards to the Marketed Reference Product
Brief Title: Bioavailability of Clotiazepam 5 mg With Regards to Reference Product
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Andromaco S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HP8810-02
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Bioequivalence
MeSH Terms: interventions — clotiazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clotiazepam Test Product (Experimental)
  Interventions: Drug: Clotiazepam 5 mg Test Product Coated Tablets
- Clotiazepam Reference Product (Active Comparator)
  Interventions: Drug: Clotiazepam 5 mg Reference Product Coated Tablets

INTERVENTIONS:
Drug: Clotiazepam 5 mg Test Product Coated Tablets — Investigational Medicinal Product
  Arms: Clotiazepam Test Product
Drug: Clotiazepam 5 mg Reference Product Coated Tablets — Rize (Trademark)
  Arms: Clotiazepam Reference Product

SUMMARY:
This Pivotal study will investigate the bioavailability in fasting women of 1 Tablet formulations containing Clotiazepam 5 mg.

The Pivotal study will be performed at a single site with 30 subjects. Participants will take 1 Tablet of the test product and reference product in 2 periods and 2 sequences (either test after reference or reference after test). There will be a washout of at least 7 days between each study period.

DETAILED DESCRIPTION:
The primary objective of the study is to investigate the relative bioavailability of

Clotiazepam of 1 tablet formulation with Clotiazepam 5 mg and to demonstrate bioequivalence of both formulations in terms of rate and extent of absorption:

* Test Product: Product manufactured by Tecnandina S.A., Ecuador.
* Reference Product: Rize [Trademark], product of Mitsubishi Tanabe Pharma, Japan.

The 90% confidence intervals for the intra-subject coefficient of variation (Test versus Reference Product) for the main pharmacokinetic parameters área under the plasma concentration-time curve from time zero to time t (AUC0-t) and from time zero to 72 hours (AUC0-72), and maximum plasma concentration (Cmax) for total Levonorgestrel and Ethinyl estradiol will be determined.

Participants will be confined in the study site for approximately 36 hours during each study period (for 12 hours pre-dosing and for 12 hours post dosing) during which pharmacokinetic (PK) blood samples will be obtained. 18 blood samples will be taken up to 24 hours after the administration in each period. Participants will return to the site to provide additional blood samples at 24 h and 34 h postdose.

The washout period between the two study periods will be at least 7 days. The samples from each participant will be analyzed with 2 methods of highperformance liquid chromatography-tandem mass spectrometry bioanalytical assays to quantify total Levonorgestrel and Ethinyl estradiol in plasma.

The safety objective is to evaluate the tolerability of both formulations in women by collecting adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant and non-breastfeeding women
* Women of childbearing age with an acceptable form of contraception during the study
* 18 to 55 years old inclusive; BMI greater than or equal to 18.51 and less than or equal to 29.99
* With results of laboratory tests, electrocardiogram and chest radiography in normal and / or negative or abnormal ranges but without clinical relevance and declared suitable for study by the doctor after the physical examination
* Capable to understand the Informed Consent Form

Exclusion Criteria:

* Study Site staff or family members
* With history of drug and/or alcohol abuse
* Smokers more tan 3 cigarettes every 7 days
* Vitamin supplements intake 7 days prior to the administration of the medications under study
* Any recent change in eating habits or physical exercise
* Using of pharmacological therapy (except over the counter medication use 7 days prior the study)
* Hypersensitivity to the study drug or other related compounds, history of serious adverse reactions or hypersensitivity to any medication
* Use, during 28 days prior to the start of the study, of medications known to alter liver enzyme activity
* Consumption of beverages or food containing grapefruit or pink grapefruit, within 7 days prior to each administration of the study medication and consumption of alcohol, caffeine or beverages or food containing xanthine 24 hours prior each administration of study medication until the last sample of each period
* History of any significant cardiovascular disease
* Acute disease that generates significant physiological changes from the start of the selection until the end of the study
* HIV, Hepatitis B and/or C positive
* Presence or history of thrombophlebitis, thrombosis or thromboembolic disorder, deep vein thrombosis, pulmonary embolism or known coagulopathy.
* Donation or loss of a significant volume (more tan 100 mL) of blood or plasma or platelets during the 3 months prior to the start of the study
* Subjects who have participated in any type of clinical study during the 3 months prior to the start of the study
* History of any gastrointestinal surgery that could affect drug absorption
* Presence of fainting history or fear to blood collection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-03-28 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
Total Clotiazepam: area under the plasma concentration-time curve from 0 to 34 hours (AUC0-34). | From intake and up to 34 hours after tablet intake.
  21 samples up to 34 hours will be taken after the administration in each period.
Total Clotiazepam: area under the plasma concentration-time curve from 0 to time t (AUC0-t). | From intake and up to 34 hours after tablet intake.
  21 samples up to 34 hours will be taken after the administration in each period.
Total Clotiazepam: Maximum plasma concentration (Cmax) | From intake and up to 34 hours after tablet intake.
  21 samples up to 34 hours will be taken after the administration in each period. The Cmax will be calculated.

SECONDARY OUTCOMES:
Total Clotiazepam: Time to achieve maximum plasma concentration (tmax) | From intake and up to 34 hours after tablet intake.
  21 samples up to 34 hours will be taken after the administration in each period. The tmax will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Innolab, Santiago, Chile